CLINICAL TRIAL: NCT01134289
Title: An Analysis of Photoplethysmographic Signal in Diagnostic Lumbar Sympathetic Block for Complex Regional Pain Syndrome
Brief Title: Analysis of Photoplethysmographic Signal in Lumbar Sympathetic Block
Acronym: park001
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Clinical Research Institute, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Seoul National Univ Hospital; H-0906-010-282 (Other: SeoulNUH)
Record Dates: First submitted 2010-05-19; First posted 2010-05-31 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Complex Regional Pain Syndrome
Keywords: complex regional pain syndrome; lumbar sympathetic blockade; photoplethysmography; diagnostic lumbar sympathetic blockade
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Bupivacaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lumbar sympathetic block (Active Comparator): Unilateral lumbar sympathetic blockade using chirocaine
  Interventions: Procedure: lumbar sympathetic block
- contralateral side (No Intervention)

INTERVENTIONS:
Procedure: lumbar sympathetic block — unilateral lumbar sympathetic block at L3 level using 0.2% chirocaine under C-arm fluoroscopy
  Other Names: 0.25% bupivacaine (Chirocaine, Abbott, Elverum, Norway); C-arm (OEC 9800 plus, GE Medical Systems, Salt Lake City, UT); Chiba needle (Cook Inc., Bloomington, IN)
  Arms: lumbar sympathetic block

SUMMARY:
This study aims to compare the alternative current and the direct current signal changes of photoplethysmography between both feet during one side lumbar sympathetic block.

The hypothesis is that signal changes occur earlier than other indices to decide whether it is successful following lumbar sympathetic block on only one-side.

ELIGIBILITY:
Inclusion Criteria:

* Physically examined for complex regional pain syndrome on lower extremity,
* Scheduled for diagnostic lumbar sympathetic blockade.

Exclusion Criteria:

* Graded as ASA 3 or higher,
* Below 18 or above 70 years of age, or
* Had any other contraindication for regional anesthesia.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Index of sympathetic block | 1 minute at intervals from baseline through end of procedure
  change of slope of signals of the alternative current and the direct current from foot
  The baseline is defined as the point of surgical drap.
  The end of procedure is decided when the temperature of foot is increased more than 2 degrees from baseline within 20 minutes after local anesthetics injection

SECONDARY OUTCOMES:
skin temperature changes | 1 minute at intervals during procedure
  foot temperature change from baseline
electrocardiogram | 1 minute at intervals from baseline through end of procedure
  heart rate variability measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul National University Hospital, Seoul, South Korea